CLINICAL TRIAL: NCT04271761
Title: A Prospective, Single-centre Evaluation of Carina Microphone Sensitivity and Maximum Stable Gain in Adult Recipients
Brief Title: Evaluation of Carina Microphone Sensitivity and Maximum Stable Gain in Adult Recipients
Acronym: CAMSEN
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: AI-5770
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Hearing Impairment
Keywords: cochlear implantation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Current adult recipients of Cochlear Carina System: Adults who are current recipients of the Cochlear Carina System. Participants will attend one scheduled visit where several acoustic measurements will be taken that do not require active participation by the participant.
  Interventions: Other: Non-interventional, post-market, pilot study of Carina Cochlear System

INTERVENTIONS:
Other: Non-interventional, post-market, pilot study of Carina Cochlear System — Several objective acoustic measurements will be performed that do not require active participation from the subject.

SUMMARY:
This investigation is a single-centre, prospective, single-arm, post-market, non-interventional, pilot clinical investigation designed to characterize microphone sensitivity and maximum stable gain of the Cochlear Carina System.

DETAILED DESCRIPTION:
The totally implanted Carina System is an active middle ear implant where all components are implanted under the skin. Placing a microphone under the skin affects its acoustic sensitivity and vibration sensitivity. Software is now available to enable non-intrusive microphone measurements in existing patients with the Carina device, through a wireless link to the implant. Detailed knowledge of the acoustic sensitivity of the implanted microphone and objectively measured maximum stable gain, and its inter-individual variability, will allow more accurate calculation of overall system performance, and thereby more accurate prediction of clinical outcomes.

Subjects will attend one scheduled study visit to be assessed; several objective acoustic measurements will be performed that do not require active participation from the subject. No data monitoring committee will be used for this clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older at the time of enrolment in the study
* Current recipient of a Cochlear Carina System.

Exclusion Criteria:

- Unwillingness or inability of the candidate to comply with all investigational requirements as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current adult recipient of a Cochlear Carina System.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Correia da Silva, MD, Principal Investigator — CUF Porto
Locations (1):
- CUF Porto Hospital, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Current Adult Recipients of Cochlear Carina System
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Current Adult Recipients of Cochlear Carina System
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Portugal | 14
Ear (Left/Right) [Count of Participants; unit: Participants]
  Left Ear | 6
  Right Ear | 8
Usage(years) [Mean (Standard Deviation); unit: years] | 3.1 (1.3)
Microphone Position [Count of Participants; unit: Participants]
  A-mastoid tip | 0
  A-B | 1
  B-posterior inferior | 1
  B-C | 0
  C-posterior mastoid | 9
  C-D | 1
  D-posterior | 1
  E-posterior superior | 0
  Unknown | 1
Type of HL, coupling [Count of Participants; unit: Participants]
  Sensorineural HL. incus | 7
  Mixed HL, stapes head | 6
  Mixed HL, "power stapes" | 1

OUTCOME MEASURES:

1. Primary Outcome: Acoustic Sensitivity of Implanted Carina Microphone
Description: The acoustic sensitivity of the implanted microphone was measured using a white noise acoustic test signal was presented from a loudspeaker, with the sound pressure level monitored with an external probe microphone positioned over the location of the implanted microphone and the signal level at the implanted microphone recorded through a wireless link to the Carina implant.
Time Frame: from date of enrolment through to study visit, an average of 1 month
Measure: Median (Full Range); unit: dB
Arm/Group | Current Adult Recipients of Cochlear Carina System
Number analyzed (Participants) | 14
dB | -64 [-95 to -53]

2. Primary Outcome: Ratio of Response of Carina Microphone : Accelerometer for Acoustic Stimulation
Description: Ratio [dB] of response of implanted microphone to response of implanted accelerometer, in-situ, for audiometric frequencies 250-6000 Hz, median and percentiles
Time Frame: from date of enrolment through to study visit, an average of 1 month
Measure: Median (Full Range); unit: MAR (Microphone : Accelerometer ratio)
Arm/Group | Current Adult Recipients of Cochlear Carina System
Number analyzed (Participants) | 14
MAR (Microphone : Accelerometer ratio) | 16.7 [-10.8 to 22.6]

3. Primary Outcome: Carina Maximum Stable Gain
Description: Transfer function from Carina output to actuator [dB FS] to Carina input from implanted microphone [dB FS], for audiometric frequencies 250-6000 Hz, with ear canal open and ear canal plugged.
Time Frame: from date of enrolment through to study visit, an average of 1 month
Measure: Median (Full Range); unit: dB
Arm/Group | Current Adult Recipients of Cochlear Carina System
Number analyzed (Participants) | 14
dB
  Ear Canal Open | 33.2 [21 to 40.7]
  Ear Canal plugged | 0.3 [-1.7 to 2.3]

4. Primary Outcome: Carina Microphone Impulse Response for Acoustic and Actuator Stimulation
Description: Identification of the system's acoustic and vibration transfer functions including non-linear components.
Time Frame: from date of enrolment through to study visit, an average of 1 month
Measure: Number; unit: participants
Arm/Group | Current Adult Recipients of Cochlear Carina System
Number analyzed (Participants) | 14
participants
  Presence of Vibration | 0
  Presence of distortion | 0

ADVERSE EVENTS:
Time Frame: There were no adverse events reported in this study. The study was a single visit and adverse events only needed to be reported from time of enrolment to completion for each subject (ie a single day).
Arm/Group | Current Adult Recipients of Cochlear Carina System
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: CIP CAMSEN AI-5770 (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT04271761/Prot_SAP_000.pdf